CLINICAL TRIAL: NCT05964257
Title: A Double-blind, Randomized, Placebo-controlled, Multi-center, Phase III Study to Evaluate the Efficacy and Safety of LIZTOX in Subjects with Benign Masseteric Hypertrophy.
Brief Title: To Evaluate the Efficacy and Safety of LIZTOX in Subjects with Benign Masseteric Hypertrophy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Huons Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HU-014_P3_BMH
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Benign Masseteric Hypertrophy
Keywords: BMH
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HU-014 (Experimental)
  Interventions: Drug: Botulinum toxin type A
- Placebo (Placebo Comparator)
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin type A(HU-014) will be administered intramuscularly to the bilateral masseter muscles on Visit 2.
  Arms: HU-014
Drug: normal Saline — Normal Saline will be administered intramuscularly to the bilateral masseter muscles on Visit 2.
  Arms: Placebo

SUMMARY:
A double-blind, randomized, placebo-controlled, multi-center, phase III study to evaluate the efficacy and safety of LIZTOX in subjects with benign Masseteric hypertrophy

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject over 19 years of age and written informed consent is obtained.
* Subject who has bilaterally symmetrical of masseter at visual and palpable assessment.
* Subject who average masseter muscle thickness of at least 14mm on each side in males and 12mm in females at maximum clenching by ultrasonography.
* Subject who has a masseter muscle hypertrophy scale of 4(marked) or more as determined by investigator.
* Subject who fully understands this clinical trial and voluntarily writes ICF in the clinical trial.

Exclusion Criteria:

* Subject who had previously received botulinum toxin within 12 weeks prior to the study entry.
* Subject who got any facial aesthetic procedure (e.g. surgery, laser, thread treatment etc.) in masseter muscle area within 48 weeks prior to the study entry.
* Subject who has a disease(e.g. Temporo mandibular joint disorder, etc.)
* Subject who were diagnosed Myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other condition that might influence with neuromuscular function.
* Subject who had taken medication(e.g. muscle relaxant, polypeptide antibiotics, aminoglycoside antibiotics, etc.) within 4 weeks prior to the study entry.
* Subject who are hypersensitive to investigational drug components (botulinum toxin, serum albumin, etc.)
* Subject who are pregnant or lactating or planing pregnancy or disagreed to avoid pregnancy during study period.
* Subject who participate other clinical trials within 4 weeks prior to the study entry.
* Subject who are not eligible for this study at the discretion of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Average change from baseline in masseter muscle thickness on both sides at maximum clenching | 12weeks
  The thickness of the masseter muscle is measured using ultrasonography, and the average value is obtained from three measurements.

SECONDARY OUTCOMES:
Average change from baseline in masseter muscle thickness on both sides at maximum clenching | 4, 8, 16, 20, 24weeks
  The thickness of the masseter muscle is measured using ultrasonography, and the average value is obtained from three measurements.
Average change from baseline in masseter muscle thickness on both sides at rest | 4, 8, 12, 16, 20, 24weeks
  The thickness of the masseter muscle is measured using ultrasonography, and the average value is obtained from three measurements.
Average rate change from baseline in masseter muscle thickness on both sides at maximum clenching | 4, 8, 12, 16, 20, 24weeks
  The thickness of the masseter muscle is measured using ultrasonography, and the average value is obtained from three measurements.
Average rate change from baseline in masseter muscle thickness on both sides at rest | 4, 8, 12, 16, 20, 24weeks
  The thickness of the masseter muscle is measured using ultrasonography, and the average value is obtained from three measurements.
Change from baseline in the lower facial volume at maximum clenching and at rest using Morpheus 3D imaging | 4, 8, 12, 16, 20, 24weeks
  When measuring, the volume of the lower face was measured twice and the average value was used.
Rate of change from baseline in the lower facial volume at maximum clenching and at rest using Morpheus 3D imaging | 4, 8, 12, 16, 20, 24weeks
  When measuring, the volume of the lower face was measured twice and the average value was used.
The proportion of subjects who reported an overall improvement of more than 50% at maximum clenching and at rest. | 4, 8, 12, 16, 20, 24weeks
  Overall improvement criteria: +4 (100% complete improvement) ~ -4 (100% very marked worsening)
The proportion of subjects who rated overall satisfaction as 'satisfied' at maximum clenching and at rest | 4, 8, 12, 16, 20, 24weeks
  Overall satisfaction criteria: grade 1 (very dissatisfied) ~ grade 7 (very satisfied), Grade 6 or higher (satisfied, very satisfied) is evaluated as satisfied.
The proportion of subjects with a masseter muscle hypertrophy scale (MMHS) ≤3 | 4, 8, 12, 16, 20, 24weeks
  MMHS Evaluation criteria: The facial contour and the condition of the bilateral masseter muscles are assessed on a scale from grade 1 (minimal) to grade 5 (very marked).

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Dongjak, Seoul, South Korea